CLINICAL TRIAL: NCT01988870
Title: A Pilot, Single Arm, Study of the Safety and Feasibility of Single-Fraction Intraoperative Radiation Treatment (IORT) With CT-On-Rails-Guided HDR Brachytherapy for the Treatment of Early-Stage Breast Cancer
Brief Title: IORT (Intra-operative Radiation Therapy) in Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shayna Showalter, MD (Other)
Responsible Party: Sponsor-Investigator, Shayna Showalter, MD, Assistant Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17091
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra-operative Radiation Therapy (IORT) (Experimental): Following breast conserving surgery, a CT-based plan will be prepared to deliver highly conformal IORT and the treatment will be administered.
  Interventions: Radiation: Intra-operative Radiation Therapy (IORT)

INTERVENTIONS:
Radiation: Intra-operative Radiation Therapy (IORT) — IORT is a form of APBI (accelerated partial breast irradiation) that allows for a high degree of dose homogeneity, exclusion of non-affected structures, and reduction of the volume of breast tissue exposed.

SUMMARY:
The purpose of this study is to evaluate an investigational way to provide radiation therapy to treat breast cancer at the time of surgery.

Traditionally, the recommended treatment for early stage breast cancer is surgery to remove the tumor, followed by whole breast radiation therapy to decrease the chance of recurrence of the cancer. Whole breast radiation involves daily radiation treatments for 4-6 weeks and can be associated with damage to other tissues including the skin. Recent technological advances have made it possible to provide radiation treatment during the breast cancer surgical procedure. This procedure is called intraoperative radiation therapy (IORT). The University of Virginia has a unique IORT system which allows for the inclusion of cutting edge imaging technology into the IORT procedure in order to provide delivery of radiation directly to the needed areas and to avoid radiation to other tissues.

ELIGIBILITY:
Inclusion Criteria:

* Women 50 years of age of older
* Patient has elected breast conserving surgical treatment for early-stage breast cancer
* Patient meets American Society for Therapeutic Radiation Oncology (ASTRO) criteria for a "suitable" or "cautionary" patient
* Life expectancy of more than 2 years
* Tumor size 4cm or less
* Women of childbearing potential must agree to use adequate contraception

Exclusion Criteria:

* Male
* Pregnant or nursing
* Any contraindication to radiotherapy
* Breast cancer that involves skin or chest wall, bilateral breast cancer or history of breast cancer in ipsilateral breast
* Patient meets any of the ASTRO criteria for an "unsuitable" patient
* Patient requires chemotherapy within two weeks of IORT
* Breast implants
* A serious uncontrolled medical disorder
* Significant history of uncontrolled cardiac disease or CNS disease

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
IORT (Intra-operative Radiation Therapy) treatment interval | 90 minutes or less
  Evaluation of the time from the acquisition of the initial CT-on-rails until the time at which IORT is complete
Overall incidence of adverse events and major toxicities | Up to 6 months following treatment

SECONDARY OUTCOMES:
IORT treatment parameters | up to 6 hours
  Gather preliminary data on planning time
Cosmetic Outcome | Up to 6 months following treatment
  Digital photographs will be taken and used to assess breast characteristics (i.e. color/pigmentation, size, shape) and evaluated for cosmetic outcomes
Quality of life assessment | Up to 6 months following treatment
  Patients will complete a breast cancer specific quality of life survey
IORT treatment parameters | upto 6 hours
  gather preliminary data on total radiation delivery time
IORT treatment parameters | upto 6 hours
  Gather preliminary data on total procedure time
IORT treatment parameters | upto 6 hours
  Gather preliminary data on dosimetry

CONTACTS AND LOCATIONS:
Overall Officials: Shayna Showalter, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States